CLINICAL TRIAL: NCT05627908
Title: Detection of Post-traumatic Abdominal Pseudoaneurysms by CEUS and CT: A Prospective Comparative Global Study
Brief Title: The PseAn Study - Study Protocol
Acronym: PseAn
Status: Recruiting | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S_09_11_21_5555
Record Dates: First submitted 2022-11-17; First posted 2022-11-28 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Abdominal Trauma; Follow-up in Abdominal Trauma
Keywords: trauma; CT scan; CEUS; follow up; abdominal pseudoaneurism
MeSH Terms: conditions — Abdominal Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- abdominal trauma: CEUS in detecting post-traumatic splenic, hepatic, and renal PAs
  Interventions: Other: Contrast-enhanced ultrasound

INTERVENTIONS:
Other: Contrast-enhanced ultrasound — Patients data monitoring with medium- and high-grade trauma to the liver, spleen, and kidney

SUMMARY:
The researchers aim to study the role of contrast ultrasound in detecting post-traumatic splenic, hepatic, and renal PAs compared with the gold standard of CT with intravenous contrast at different follow-up time points, and whether it can replace CT scan in the follow-up of solid organ injuries

DETAILED DESCRIPTION:
Adult patients (18 years old and above) with proven blunt or penetrating splenic and/or liver and/or renal trauma as shown by a CT scan and classified according to the American Injury Scale American Association for Surgery (AAST) Organ Injury Scale (OIS) with OIS III and above will undergo a follow-up with both a CEUS and CT scan to detect post-traumatic parenchymal pseudoaneurysm within two to five days from injury. Follow-up over five days post-admission will be included if they were performed within the same hospitalization

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18 years old and above) with proven blunt or penetrating splenic and/or liver and/or renal trauma as shown by a CT scan and classified according to the American Injury Scale American Association for Surgery (AAST) Organ Injury Scale (OIS) will be included

Exclusion Criteria:

* minor to 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients (18 years old and above) with proven blunt or penetrating splenic and/or liver and/or renal trauma as shown by a CT scan and classified according to the American Injury Scale American Association for Surgery (AAST) Organ Injury Scale (OIS) will be included
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pseudoaneursim (PA) | up to 5 days post patients admission
  In each centre, the coordinator will collect epidemiological, clinical, and surgical data on a case report form (CRF) that will be completed through a questionnaire by accessing a protected database.
  The protocol for data collection is shown in appendix 1 (attached). The link for accessing the completion of the CRF will be sent by email, to the Main Lead of each participating centre.
  The main outcome will be the number of post-traumatic Pseudoaneurysms identified with CT scan and CEUS.
  The sample size for unknown populations has been derived according to the formula N= Z2 x p (1-p)/ e2, setting standard deviation (SD) at 50%, confidence interval at 95%, and Z-score at 1.65. The minimum sample size was 385 patients with a sampling error of ± 5%.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No